CLINICAL TRIAL: NCT02916966
Title: Case-control and Population Questionnaire Studying Environmental Risk Factors and Neurological Diseases
Brief Title: Environmental Exposure and Neurological Diseases Questionnaire
Acronym: Cleveland Ohio
Status: Completed | Type: Observational
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Elijah W. Stommel, Professor of Neurology, Dartmouth-Hitchcock Medical Center
Other Study IDs: D06019
Record Dates: First submitted 2016-09-26; First posted 2016-09-28 (Estimated); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (4):
- ALS Patients in Case-Control: ALS patients enrolled by Cleveland Clinic Foundation (CCF)
  Interventions: Other: Patient Registry
- Non-neurodegenerative patients in case control: Non-neurodegenerative patients enrolled by CCF
  Interventions: Other: Patient Registry
- Non-neurodegeneration population in population control: Non-neurodegenerative general population enrolled by ABS mailing system from DHMC
  Interventions: Other: Patient Registry
- ALS Patients in State of OH: ALS registry of all cases in Ohio
  Interventions: Other: Patient Registry

INTERVENTIONS:
Other: Patient Registry — Patient Registry

SUMMARY:
The proposed research is particularly relevant to the National ALS Registry and public environmental health issues because it addresses the potential environmental causes of sporadic ALS. The research will develop an ALS surveillance program in Ohio that can be compared with the national and State-Metro Surveillance Programs of the National ALS Registry, and novel methodologies to determine the role of the cyanobacterial toxin, BMAA (beta-methylamino-L-alanine), and other environmental toxins/toxicants as risk factors for ALS. This work will advance the mission of the Centers for Disease Control Agency for Toxic Substances and Disease Registry (CDC ATSDR) National ALS Registry by offering data on ALS cases in Ohio that address public health concerns over the effects of chronic exposure to cyanobacterial blooms in Lake Erie.

ELIGIBILITY:
Inclusion Criteria:

* ALS
* Non-neurodegenerative controls
* Can willingly give consent
* Over 18 years of age

Exclusion Criteria:

* Cannot give consent
* Under 18 years of age

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. ALS patients in case-control at CCF
  2. Non-neurodegenerative patients in case control at CCF
  3. Non-neurodegenerative general population in Ohio
  4. ALS patient registry in Ohio
Sampling Method: Probability Sample
Enrollment: 460 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2023-09 (Actual); Study Completion 2023-09 (Actual)

PRIMARY OUTCOMES:
Questionnaire for Environmental Exposures, Toxins, and Neurological Disease | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States